CLINICAL TRIAL: NCT05470517
Title: Antibiotic Instillation in Acute Complex Appendicitis for Prevention of Deep Space Surgical Site Infections
Brief Title: Antibiotic Instillation in Appendicitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00323208
Record Dates: First submitted 2022-07-19; First posted 2022-07-22 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Complicated Appendicitis; Acute Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Ceftriaxone

STUDY DESIGN:
Intervention Model Description: Single-blinded randomized controlled pilot phase 2 study
Who Masked: Participant
Masking Description: The surgeon and team administering the treatment will not be blinded; however, patients, patients' families, and hospital caregivers outside of the operating room will be blinded to the treatment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Arm A) (Active Comparator): Intra-operative aspiration of intra-peritoneal fluid after successful appendectomy.
  Interventions: Procedure: Intra-peritoneal Fluid Aspiration
- Standard of Care and Antibiotic instillation (Arm B) (Experimental): Intra-operative aspiration of intra-peritoneal fluid after successful appendectomy and subsequent instillation of 10ml of intra-peritoneal ceftriaxone (2g)
  Interventions: Drug: Ceftriaxone; Procedure: Intra-peritoneal Fluid Aspiration

INTERVENTIONS:
Drug: Ceftriaxone — Ceftriaxone is a sterile, semisynthetic, broad-spectrum cephalosporin antibiotic for intravenous, intramuscular, or intra-peritoneal administration.
  Ceftriaxone is a white powder, which is soluble in water. In this study ceftriaxone crystalline powder will be dissolved in 0.9% sodium chloride solution prior to intra-peritoneal instillation.
  Antibiotic instillation will be introduced into the RLQ/pelvis after the appendectomy is completed and all intra-peritoneal fluid is aspirated. Ceftriaxone solution will be used depending on availability and pharmacy stock for use at Johns Hopkins All Children's Hospital. The ceftriaxone powder (2g) will be dissolved in 9ml of sterile normal saline, for a total instillation volume of 10ml. This fluid will then be instilled and left to dwell in the area of the peritoneal cavity where the appendix was removed.
  Other Names: Ceftriaxone sodium
  Arms: Standard of Care and Antibiotic instillation (Arm B)
Procedure: Intra-peritoneal Fluid Aspiration — Intra-operative aspiration of intra-peritoneal fluid after successful appendectomy.

SUMMARY:
Appendicitis (inflammation of the wall of the appendix, causing pain and tenderness in the abdomen) has a range of severity that goes from simple to complicated. Complicated appendicitis may present with infected fluid inside of the abdomen or a perforation or hole in the intestines.

This research is being done to determine if placing an antibiotic solution in the abdomen at the time the appendix is removed is a safe procedure in patients between the ages of 3 and 18 years old with findings of complicated appendicitis.

Johns Hopkins All Children's Hospital (JHACH)'s current standard of care for patients with complicated appendicitis includes suctioning the infected fluid out of the abdomen at the time the appendix is removed. As part of this study, the investigators would like to see if patients with complicated appendicitis will benefit from routine care plus leaving an antibiotic solution inside the abdomen, after fully suctioning the infected fluid out of the abdomen.

DETAILED DESCRIPTION:
Appendicitis is one of the most common surgical diagnoses in the pediatric population and the most common surgical emergency in children. In complex appendicitis, the sequelae have progressed beyond the confines of the organ, and have led to purulent fluid in the intra-abdominal space, spillage of intestinal contents, or gross perforation of the appendix. Complicated appendicitis occurs in up to 20% of cases and is associated with a much higher morbidity and mortality. Previous studies have shown that local treatment of peritonitis associated with peritoneal dialysis (PD) catheters with intra-peritoneal antibiotics has had significant improvement of outcomes. The intra-peritoneal route is preferable as compared to oral and intravenous antibiotic administration due to elevated local levels of the antibiotic above the minimum inhibitory concentration while avoiding venipuncture and systemic side effects. There is minimal risk associated with involvement in this study given that the investigators will be screening for any history of allergies to penicillin or cephalosporins, and excluding these patients. Ceftriaxone is commercially available, has a low risk profile, and is generally well tolerated with minimal side effects.

The investigators' treatment period will include a one-time intra-operative dose of intra-peritoneal ceftriaxone (or an appropriate second or third generation cephalosporin to be designated at the discretion of the institutional Antibiotic Stewardship committee should ceftriaxone be unavailable). Typical dosing strategies for intra-peritoneal ceftriaxone administration occur on a daily basis, so the investigators' treatment period will also include the 24 hours following intra-peritoneal administration of ceftriaxone. All patients diagnosed with acute complicated appendicitis intra-operatively, and entered into the investigators' study, will also receive a minimum 48 hours of intravenous antibiotics as an inpatient, allowing for continued observation. The investigators will be treating pediatric patients who are intra-operatively diagnosed with complex appendicitis, as defined by any of the following: visible hole in the appendix, extra-luminal fecalith, diffuse fibropurulent exudate outside the right lower quadrant (RLQ)/pelvis, or intraperitoneal abscess. All patients will have been admitted to Johns Hopkins All Children's Hospital with a diagnosis of acute appendicitis prior to surgical intervention. Patients will then be randomized once diagnosed with complex appendicitis intra-operatively. Patients with allergies to penicillin or cephalosporins will be excluded pre-operatively, as well as patients who do not meet the weight requirement, are pregnant, being treated non-operatively, and those who have been intra-operatively diagnosed with simple appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute appendicitis and are scheduled to undergo urgent appendectomy
* Between 3-18 years of age at time of appendectomy
* Has intraoperative findings of complex appendicitis defined by: visible hole in the appendix, extra-luminal fecalith, diffuse fibropurulent exudate outside the RLQ/pelvis, or intraperitoneal abscess
* Weighs equal to or greater than 20kg at time of surgery

Exclusion Criteria:

* Pregnant
* Has a penicillin or cephalosporin allergy that is severe or anaphylactic in nature, prohibiting the use of these antibiotics
* Has simple appendicitis
* Undergoes appendectomy following failed or planned medical management of appendicitis
* Has impaired renal function (CrCl <15mL/min)
* Has history of neurological conditions such as encephalopathy, seizures, myoclonus and non-convulsive status epilepticus
* Has a known inability to complete a 30-day postoperative follow up

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 190 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole M. Chandler, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Those eligible preoperatively (n=337) were approached for consent with the caveat that they are eligible intraoperatively (complicated appendicitis). The number of patients who were consented (190) is not the same as the number of patients who were randomized (32). The remaining 158 eligible participants were not randomized due to intraoperative findings (n=156) and screen failures (n=2).
Groups:
- Standard of Care and Antibiotic Instillation (Arm B): Intra-operative aspiration of intra-peritoneal fluid after successful appendectomy and subsequent instillation of 10ml of intra-peritoneal ceftriaxone (2g)
  Ceftriaxone: Ceftriaxone is a sterile, semisynthetic, broad-spectrum cephalosporin antibiotic for intravenous, intramuscular, or intra-peritoneal administration.
  Ceftriaxone is a white powder, which is soluble in water. In this study ceftriaxone crystalline powder will be dissolved in 0.9% sodium chloride solution prior to intra-peritoneal instillation.
  Antibiotic instillation will be introduced into the RLQ/pelvis after the appendectomy is completed and all intra-peritoneal fluid is aspirated. Ceftriaxone solution will be used depending on availability and pharmacy stock for use at Johns Hopkins All Children's Hospital. The ceftriaxone powder (2g) will be dissolved in 9ml of sterile normal saline, for a total instillation volume of 10ml. This fluid will then be instilled and left to dwell in the area of the peritoneal cavity where the appendix was removed.
  Intra-peritoneal Fluid Aspiration: Intra-operative aspiration of intra-peritoneal fluid after successful appendectomy.
Period: Overall Study
Arm/Group | Standard of Care (Arm A) | Standard of Care and Antibiotic Instillation (Arm B)
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (Arm A) | Standard of Care and Antibiotic Instillation (Arm B) | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.96 (3.77) | 11.58 (3.96) | 11.77 (3.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 9 | 12 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Use of Antibiotic Solution Instillation Following Intraoperative Diagnosis of Complex Appendicitis as Assessed by Percentage of Eligible Participants Who Agree to Participate
Description: The study will be deemed feasible if >50% of potential participants agree to participate. This benchmark is based on a previous similar study completed in this population.
Time Frame: Up to 30 days postoperatively
Population: Patients With Appendicitis Eligible for Study
Measure: Count of Participants; unit: Participants
Groups:
- Number of Patients With Appendicitis Eligible for Study: Patients between the ages of 3 and 18 years old who present with acute appendicitis that will be managed with operative intervention.
Arm/Group | Number of Patients With Appendicitis Eligible for Study
Number analyzed (Participants) | 337
Participants
  Number of Patients Eligible who Declined Study Participation | 147
  Total number of Eligible Patients who Agreed to Participate | 190

2. Primary Outcome: Feasibility of the Use of Antibiotic Solution Instillation Following Intraoperative Diagnosis of Complex Appendicitis as Assessed by Percentage of Randomized Participants Who Complete All Intervention Sessions and Measurement Time Points
Description: The study will be deemed feasible if at least 75% of randomized participants complete all intervention sessions and measurement time points per study protocol. This benchmark is based on a previous similar study completed in this population.
Time Frame: Up to 30 days postoperatively
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care (Arm A) | Standard of Care and Antibiotic Instillation (Arm B)
Number analyzed (Participants) | 16 | 16
percentage of participants | 100 | 81

3. Primary Outcome: Safety of the Use of Antibiotic Solution Instillation Following Intraoperative Diagnosis of Complex Appendicitis as Assessed by Number of Adverse Events
Description: Safety will be determined by adverse events in all participants.
Time Frame: Up to 30 days postoperatively
Measure: Number; unit: adverse events
Arm/Group | Standard of Care (Arm A) | Standard of Care and Antibiotic Instillation (Arm B)
Number analyzed (Participants) | 16 | 16
adverse events | 11 | 17

ADVERSE EVENTS:
Time Frame: Up to 30 days post operatively
Arm/Group | Standard of Care (Arm A) | Standard of Care and Antibiotic Instillation (Arm B)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 9/16 | 8/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (Arm A) (N=16) | Standard of Care and Antibiotic Instillation (Arm B) (N=16)
laparotomy, lysis of adhesions, omenectomy (Surgical and medical procedures) | 0 (0) | 1 (1) — 1. Single incision diagnostic laparotomy 2. Exploratory laparotomy with lysis of adhesions 3. Omentectomy 4. Incisional negative pressure wound therapy
post-op skin redness/blotches (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
abscess/fluid collection (Infections and infestations) | 7 (7) | 4 (5)
non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
bladder infection (Infections and infestations) | 0 (0) | 1 (1)
drain exchange/placement (Surgical and medical procedures) | 0 (0) | 1 (2)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) — grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/17/NCT05470517/Prot_SAP_000.pdf